CLINICAL TRIAL: NCT03094767
Title: Cardiorespiratory Parameters and Glycated Hemoglobin of Patients With Type 2 Diabetes After a Rehabilitation Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: União Educacional do Norte (Other)
Responsible Party: Principal Investigator, NATÁLIA DA SILVA FREITAS MARQUES, Principal Investigator, Clinical Research, União Educacional do Norte
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1.616.721
Record Dates: First submitted 2017-02-25; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2; Rehabilitation; Respiratory Therapy
Keywords: Type 2 Diabetes Mellitus; Heart Rate Variability; Rehabilitation; Hemoglobin Glycated
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Experimental): Patients will be submitted only to the initial protocol of rehabilitation, i. e., they will have only one session on the initial day and one session on the final day, after 12 weeks.
  Interventions: Other: Initial and Final assessment
- Interventional Group (Experimental): Patients will participate in the cardiovascular rehabilitation program during 12 weeks.
  Interventions: Other: Cardiovascular Rehabilitation; Other: Initial and Final assessment

INTERVENTIONS:
Other: Cardiovascular Rehabilitation — Aerobic and anaerobic exercises performed for 12 weeks, 3x/week, of 60 minutes each.
  Arms: Interventional Group
Other: Initial and Final assessment — Measuring blood preassure, heart rate, Borg scale, respiratory rate, oxygen saturation and HbA1C in the first day of assessment and after 12 weeks.

SUMMARY:
Cardiovascular autonomic dysfunction reflects the pathophysiology of Diabetes Mellitus in this patient group favors an increase in morbidity and mortality related to cardiovascular events, and for this reason has been one of the most studied clinical entities.

Therefore this work aims to analyze the cardiorespiratory parameters and glycated hemoglobin after the commission of a rehabilitation program in patients with diabetes mellitus type 2.

The collection protocol is to check the heart rate, blood pressure, double product, Borg scale, variability heart rate and glycated hemoglobin of patients with type 2 diabetes This project this is an experimental study, the type randomized clinical trial on the hemodynamic response and glucose levels in patients with DM2 institutionalized in Acre Hospital Foundation submitted to one rehabilitation program consisting of aerobic and anaerobic exercises performed for 12 weeks in three weekly meetings, of 60 minutes each.

DETAILED DESCRIPTION:
Background: Built with evidence that makes it possible to work in cardiac rehabilitation programs in patients with type 2 diabetes with more security, guaranteeing them an improvement in cardiorespiratory fitness, the hemodynamic and glycemic variables, allowing them a better quality of life

Method/Design: The research instrument is applied before and after the practice of the proposed exercise program (consisting of aerobic and anaerobic exercises performed for 12 weeks in three weekly meetings, of 60 minutes each). The instrument is based on the following collection protocol: assessment of BP, HR, Borg scale, respiratory rate (RR), oxygen saturation (SAT), the DP calculation and will be carried out the examination to check HbA1C Will be performed for 12 weeks in three weekly meetings, of 60minutes each, in total of 36 sessions with antecipated 60 pacients splited in 2 groups "Control" and "intervention"

Discussion: Correlate the variability of heart rate behavior and glycated hemoglobin after the exercise program; To demonstrate the possible association between the change of the cardiorespiratory parameters according to the variation of glycated hemoglobin; Demonstrate the possibility of association between the variation of the cardiorespiratory parameters and glycated hemoglobin according to sex;

ELIGIBILITY:
Inclusion Criteria:

* type 2 Diabetes
* Sedentary
* Non-smoker
* with medical prescription for rehabilitation program.

Exclusion Criteria:

* Neurological disease
* Acute heart failure
* Morbid obesity
* Atrial fibrillation
* Sick sinus syndrome
* Atrioventricular block grade II or III
* Who used beta-blockers
* Who used antiarrhythmic medication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Heart rate variability at 3 months | three months
  With a specific heart rate monitor, Heart Rate Variability (also called RR variability) is the measure of heart rate variation between each pair of heart beats at a given time interval.
  The results of the heart rate variability analysis are divided into two groups: time domain results and frequency domain results.
  They are numbers related to the "rhythm" in which the variations occur:
  VLF - Very Low Frequency: power contained in the range below 0.04Hz. LF - Low Frequency: power contained in the range of 0.04 to 0.15Hz. HF - High Frequency: power contained in the range of 0.15 to 0.4Hz. LF / HF: Ratio between LF and HF powers.
Change from baseline of Glycated Hemoglobin at 3 months | three months
  The HbA1c test counts the number of red blood cells that are glycated, that is, linked to a glucose molecule.

SECONDARY OUTCOMES:
Change from baseline of pulse oximetry at every intervention session | three months
  With the use of pulse oximetry we will observe the percentage of oxygen that the blood is carrying, compared to the maximum of its transport capacity. Ideally, more than 89% of your red cells should be carrying oxygen.
Change from baseline of subjective sensation of respiratory discomfort at every intervention session | three months
  Used on the modified borg scale cr 410 that goes with a score of 0 to 10 where the patient will identify their degree of discomfort after the protocol in which it was submitted;
Change from baseline of Blood Pressure at every intervention session | three months
  The expression blood pressure (BP) or blood pressure refers to the pressure exerted by the blood against the wall of the arteries. Blood pressure as well as that of the whole circulatory system is usually slightly above atmospheric pressure, the pressure difference being responsible for keeping the arteries and other vessels not collapsed. In a healthy person, the amount of pressure can vary continuously, depending on the stress, the emotion or if you are doing physical activity.
Change from baseline of the distance traveled at 3 months. | three months
  This will be measured in meters during a six-minute walk test in a 30-meter runner where the participant should walk as mush as he/she can in six minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia da Silva Freitas Marques, Master, Principal Investigator — União Educacional do Norte
Locations (1):
- União Educacional do Norte, Rio Branco, Acre, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marques NDSF, Abreu LC, Santos BVD, Neto CFR, Silva JRCD, Braga KKS, Uchoa KDS, Moraes LMS, Ferreira LCP, Ribeiro NG, Santos SLD, Silva TAD, Andrade PE, Raimundo RD. Cardiorespiratory parameters and glycated hemoglobin of patients with type 2 diabetes after a rehabilitation program. Medicine (Baltimore). 2018 Feb;97(8):e9321. doi: 10.1097/MD.0000000000009321. PMID 29465549